CLINICAL TRIAL: NCT06973811
Title: A Prospective, Phase II Clinical Trial Using the Combination of Zanubrutinib, Rituximab and High-dose Intravenous Methotrexate With Intravitreal Methotrexate Injection Therapy for the Treatment of Primary Intraocular Lymphoma
Brief Title: ZR-MTX for PIOL Phase II Trial
Acronym: ZR-MTX
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhang, Prof., Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K6396
Record Dates: First submitted 2025-05-06; First posted 2025-05-15 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Primary Intraocular Lymphoma
Keywords: primary intraocular lymphoma
MeSH Terms: conditions — Intraocular Lymphoma | interventions — Methotrexate; Rituximab; zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZRMTX (Experimental): Zanubrutinib/Rituximab/IV MTX & intravitreal MTX Experimental arm will be treated with rituximab plus zanubrutinib (ZR) regimen for 4 cycles, ZR plus iv MTX for 2 cytles and followed by zanubrutinib maintenance for 2 years ( or choose to stop zanubrutinib maintenance if reached CR with negative CSF cfDNA). Meanwhile, intravitreal methotrexate will be given as protocol during the 1st year of treatment.
  Interventions: Drug: Methotrexate; Drug: Rituximab (R); Drug: Zanubrutinib; Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Methotrexate — 400ug intravitreal injection every week for 4 doses in the induction phase, every 2 weeks for 2 doses as consolidation, then every month for 10 doses
Drug: Rituximab (R) — Rituximab 375mg/m2 intravenous infusion d1, every 21 days for 1 cycle. 6 cycles will be prescribed as protocol
Drug: Zanubrutinib — 160mg Bid, oral. 21-day cycle for 6 cycles in the induction phase and for 2 years in the maintenance phase
Drug: Methotrexate (MTX) — Methotrexate 3.5g/m2 intravenous infusion d1, every 21 days for cycle 5 and 6 only.

SUMMARY:
This is a prospective single-arm phase II study, with the purpose of evaluating the efficiency of ZR-MTX regimen (Rituximab, Zanubrutinib and methotrexate) combined with intravitreal methotrexate, then followed by minimal residual disease directed Zanubrutinib maintenance in newly-diagnosed primary intraocular lymphoma. The primary endpoint of this study is progression-free survival (PFS).

DETAILED DESCRIPTION:
All the patients will be treated with ZR regimen (Rituximab 375mg/m2 IV d1, Zanubrutinib 160mg Bid, 21 days per cycle) as induction regimen. The response will be evaluated after 2 cycles of ZR regimen. Patients who achieved complete remission (CR) or partial remission (PR) or stable disease (SD) will receive 2 more cycles of ZR regimen. The patients with progressed disease (PD) will withdraw from the trial and receive salvage regimens. Then 2 more cycle of ZR regimen will be administrated. Patients will be evaluated again, those achieved CR or PR or SD will continue to receive 2 cycles of ZR-MTX regimen (Rituximab 375mg/m2 IV d1, Methotrexate 3.5g/m2 IV d1, Zanubrutinib 160mg Bid, 21 days per cycle), while those PD will drop out. In the meantime, intravitreal methotrexate will be given at a dose of 400ug for 16 doses. After total 6 induction cycles, the investigators evaluate the efficiency again, the patients with CR and MRD negativity (by CSF IL-10 and cfDNA) will stop treatment. Those with MRD positive CR or PR or SD will go to Zanubrutinib maintenance for 2 years or until progression of the disease (PD), unacceptable toxicity, or patient/investigator discretion. And the patients with PD will receive a salvage regimen. During following-up, surveillance ophthalmologic examination, and brain magnetic resonance imaging (MRI) scans can be performed every 3 months up to the first 2 years, followed by the doctor's visit every 6 months for up to 5 years or disease relapses.

ELIGIBILITY:
Inclusion Criteria:

* • Newly-diagnosed primary vitreoretinal lymphoma

  * ECOG≤2
  * creatinine clearance rate (CCR) ≥ 60ml/h, according to Cockcroft-Gault
  * Total bilirubin # 2 upper limits of normal, alanine aminotransferase#ALT# < 3 upper limits of normal
  * Sign the Informed consent
  * Women of childbearing potential must understand that the study medication could have a potential teratogenic risk. They should undergo complete contraception during the study period.
  * Male subjects must agree to use condoms throughout study drug therapy.

Exclusion Criteria:

* • primary central nervous system lymphoma involved eyes and brain

  * systemic B cell lymphoma involved eyes
  * Pre-existing uncontrolled active infection
  * Clinical evidence of grade 3 or 4 heart failure as defined by the New York Heart Association criteria
  * Pregnancy or active lactation
  * Co-existing tumors
  * HIV or HBV or HCV infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
2 years progression-free survival | from the date of treatment to the subject finished his 2 years follow-up phase or the disease relapsed or the death due to lymphoma
  2 years progression-free survival was calculated from the date of therapy until death from lymphoma or 2-year follow up without relapsing

SECONDARY OUTCOMES:
overall response rate (ORR) | 4 weeks after the end of 6 cycles of induction (each cycle is 21 days).
  ORR was calculated by the proportion of patients who achieved complete remission and partial remission.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Site demands.